CLINICAL TRIAL: NCT04907435
Title: Comparison of Simultaneous Laparoscopic and Open Operations for Synchronous Liver Metastases With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Institution Russian Scientific Center of Roentgenoradiology of the Ministry (Other)
Responsible Party: Principal Investigator, Ivanova Olga, doctor, Federal State Budgetary Institution Russian Scientific Center of Roentgenoradiology of the Ministry
Other Study IDs: 1
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Optimization of Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with simultaneous laparoscopic operations
  Interventions: Procedure: simultaneous operations
- patient with simultaneous open operations
  Interventions: Procedure: simultaneous operations

INTERVENTIONS:
Procedure: simultaneous operations — simultaneous operations

SUMMARY:
retrospective analysis of medical records of patients with synchronous liver metastatic colorectal cancer, who underwent simultaneous operations on the intestine and on the liver, from January 2011 to November 2020 at the Russian Scientific Center for Roentgenoradiology. 2 groups of 21 patients each were formed: group 1 included a patient with simultaneous laparoscopic operations, group 2 included a patient with simultaneous open operations.

ELIGIBILITY:
Inclusion Criteria:

* patients with synchronous metastatic liver lesions with colorectal cancer

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with synchronous metastatic liver lesions with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | three years

IPD SHARING:
Plan to Share IPD: No